CLINICAL TRIAL: NCT06366334
Title: A Double Blinded, Randomized, Placebo Controlled, Parallel Arm Pilot Trial of Intravenous Ketamine for Emergency Department Treatment of Suicidal Ideation in a Pediatric Population.
Brief Title: Study of IV Ketamine for Emergency Department Treatment of Adolescent Suicidal Ideation
Acronym: KSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Maala Bhatt, Associate Professor of Pediatrics, Director of Emergency Research, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23/02E
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Suicidal Ideation; Suicidal Ideas
MeSH Terms: conditions — Suicidal Ideation | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Participants in the intervention group will receive 0.5mg/kg of 1mg/mL intravenous ketamine (50 mg maximum) over 40 minutes.
  Interventions: Drug: Ketamine Hydrochloride
- Normal Saline (Placebo Comparator): Participants in the control group will receive 0.5mL/kg intravenous normal saline (50 ml maximum) over 40 minutes
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride — See arm description
  Other Names: Ketamine
  Arms: Ketamine
Drug: Normal saline — See arm description
  Arms: Normal Saline

SUMMARY:
Approximately 20% of Canadian adolescents experience thoughts of suicide, or suicidal ideation (SI), and suicide is the second leading cause of death among Canadians aged 15-19 years. The emergency department at CHEO sees approximately four patients per day with SI. Even though this is a medical emergency, there are no fast-acting treatments available.

Ketamine is a medication that is commonly used to safely sedate children who require painful procedures in the emergency department. For nearly ten years, intravenous ketamine has also been shown to rapidly reduce SI in adults. However, ketamine as a treatment for SI has never been studied in adolescents. The primary study objective is to pilot a clinical trial that investigates intravenous ketamine to emergently treat SI in adolescents.

If intravenous ketamine can relieve symptoms of SI for youth, this would have tremendous effects on patients and would dramatically change how physicians treat adolescent mental health emergencies. If ketamine is effective for several weeks, as it is in adults, it will help temporize patients until they receive more long-term psychiatric care. At the system level, it has the potential to reduce emergency visits and lengthy admissions. The investigators feel that the results of this study will be generalizable to pediatric centres across Canada and beyond.

DETAILED DESCRIPTION:
Suicidal ideation (SI) is a common and often severe cause of morbidity in adolescents. Patients frequently present to the emergency department (ED) with severe and distressing thoughts of self-harm or suicide, and yet, there is currently no acute therapeutic intervention to offer them. The standard of care for patients who do not require admission is to discharge them home with resources for websites, apps, or telephone help lines. These interactions fail to address the underlying suicidal thoughts and leave patients, families and providers feeling very dissatisfied. Medications are nearly never initiated in the ED and patients who are already taking anti-depressants experience a very slow therapeutic onset, and often with unfavourable side effects that make medication compliance difficult and sometimes impossible.

For nearly ten years, intravenous ketamine has been shown to be an efficacious acute therapy in adult patients with suicidal ideation. A single dose of intravenous (IV) ketamine can rapidly reduce the severity of suicidal ideation by moderate to large effect sizes (Cohen's d = 0.5-0.8) during an ED visit, in an adult population. However, it has never been studied in a pediatric population. The study primary objective is to determine the feasibility of conducting a trial that investigates the efficacy of IV ketamine to reduce suicidal ideation in adolescents in the pediatric emergency department.

If intravenous ketamine can rapidly alleviate the severity of SI for adolescents, this would have tremendous effects on patients and families and dramatically change how ED physicians treat pediatric mental health emergencies. It would increase patient safety, reduce patient distress, morbidity, possibly mortality and alleviate family stress. If the therapeutic effect of ketamine is maintained for several days, as it is in adults, it will help temporize patient symptoms while they are connected with more long-term psychiatric care. At the system level, it may reduce rates of ED visits and, often lengthy, admissions to hospital. The investigators feel that the results of this study will be generalizable to pediatric centres across Ontario, Canada and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. Responds "yes" to Ask Suicide Screening Question (ASQ) #5 at triage, which asks; "Are you having thoughts of killing yourself right now?"
2. Moderate to severe suicidal ideation, defined as score ≥ 3 on the first 5 questions of the Beck Scale for Suicidal Ideation (SSI5)
3. Age 12 to 17 years, inclusive
4. Medically clear (deemed fit for participation in the trial), as judged by the treating physician. Minimum criteria required to be deemed medically clear are: a) No evidence of serious physical injury requiring urgent intervention b) No evidence of acute ingestion requiring monitoring, blood tests, imaging or ECG or in the context of acute ingestion they have satisfied the requisite number of hours of post-ingestion monitoring with no further need for intervention.

Exclusion Criteria:

1. Acute intoxication from any substance, including alcohol
2. Previously enrolled in the current study or currently enrolled in another clinical trial
3. History of intellectual disability or autism spectrum disorder by patient/parent report
4. Active, or history of, psychosis or psychotic disorder
5. History of non-psychiatric neurologic disorder (e.g., epilepsy)
6. Any of the following contraindications to ketamine based on the drug monograph: a) Known allergy or hypersensitivity to ketamine by patient history b) History of cerebrovascular accident (stroke or aneurysm) c) History of elevated intracranial pressure or idiopathic intracranial hypertension d) Significant hypertension requiring daily medication e) Severe cardiac decompensation
7. On an involuntary psychiatric hold
8. Requires physical or chemical restraint
9. History of violence while in hospital
10. Pregnant or breastfeeding
11. Received opioids in the 2-hours prior to study screening

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible participants who complete the study protocol | Baseline
  This is a feasibility measure; the investigators will report the number of patients who are screened for participation, are eligible, eligible and consent, complete the intervention, complete study follow-up

SECONDARY OUTCOMES:
Baseline distribution of responses to the first 5 questions of Beck Scale for Suicidal Ideation (SSI5) | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the SSI5 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Baseline distribution of responses to the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MADRS10) | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the MADRS10 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Baseline distribution of responses to the suicide item (#9) from the Beck Depression Index (BDI9). | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the BDI9 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Baseline pragmatic assessment of the first 5 questions of the Beck Scale for Suicidal Ideation (SSI5), the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MADRS10), and the suicide item (#9) from the Beck Depression Index (BDI9). | Baseline
  Pragmatic assessment of the tool validity by asking each participant, which of the three tools best captures how they are feeling at baseline.
Assessment of blinding | Baseline
  Blinding adequacy will be measured by asking each participant which intervention they think they received at the end of the 40 minute study drug infusion.
Treatment efficacy measured by the Beck Scale for Suicidal Ideation (SSI5) | 40 minutes after the beginning of the infusion
  Change in suicidal ideation severity from baseline at the end of the 40-minute medication infusion will be measured using SSI5.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MADRS10) | 40 minutes after the beginning of the infusion
  Change in suicidal ideation severity from baseline at the end of the 40-minute medication infusion will be measured using MADRS10.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#9) from the Beck Depression Index (BDI9) | 40 minutes after the beginning of the infusion
  Change in suicidal ideation severity from baseline at the end of the 40-minute medication infusion will be measured using BDI9.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Treatment durability measured by the Beck Scale for Suicidal Ideation (SSI5) | 40, 80, 120 minutes after the beginning of the infusion as well as 24 hours and 7 days post enrollment
  The durability of a treatment effect on suicidal ideation will be measured by SSI5 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Treatment durability measured by the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MADRS10) | 40, 80, 120 minutes after the beginning of the infusion as well as 24 hours and 7 days post enrollment
  The durability of a treatment effect on suicidal ideation will be measured by MADRS10 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#9) from the Beck Depression Index (BDI9) | 40, 80, 120 minutes after the beginning of the infusion as well as 24 hours and 7 days post enrollment
  The durability of a treatment effect on suicidal ideation will be measured by BDI9 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Admission to Hospital | Enrollment visit
  Proportion of patients who require hospital admission at the enrolment ED visit
Length of Stay in Hospital | 30 days post enrollment
  The mean and standard deviation of length of hospital stay for patients admitted at the enrollment visit
ED revisits | 30-days post enrollment
  Proportion of patients who have an ED visit(s) for mental health complaints within 30 days following enrolment

OTHER OUTCOMES:
Safety Outcome 1: Clinically significant tachycardia | Enrollment visit
  Present at 120 minutes post infusion and requires intervention by the treating team
Safety Outcome 2: Clinically significant hypertension | Enrollment visit
  Present at 120 minutes post infusion and requires intervention by the treating team
Safety Outcome 3: Vomiting | Enrollment visit
  Vomiting during or after the infusion
Safety Outcome 4: Dissociation | During the infusion
  Clinician-Administered Dissociative States Scale (CADSS; minimum score 0, maximum score 24) - total score of 6 or more OR 4 on any single question AND clinically dissociated
Safety Outcome 5: Death | 30-days post enrolment
  Death from any cause within 30 days following enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Tyrus Crawford, BA, Study Director — CHEO
Locations (1):
- Children's Hospital Of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No